CLINICAL TRIAL: NCT06834113
Title: Impact of Two Types of Interventions (Ventrogluteal Versus Dorsogluteal Injection Site; Virtual Reality Headset: Presence or Absence) on Pain After Injections of Vocabria® (Cabotegravir) and Rekambys® (Rilpivirine) in Patients Infected With Human Immunodeficiency Virus -1
Brief Title: Impact of Pain From Injectables Antiretroviral Treatments in HIV-1 Patients Based on the Injection Site (Ventrogluteal or Dorsogluteal) and the Use or Non-use of Virtual Reality Headset
Acronym: VIHINJECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CHUO-2024-15
Record Dates: First submitted 2025-01-31; First posted 2025-02-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: HIV I Infection; Injection Pain

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, open-label study with a cross-over design. Eeach participant will serve as their own control and will randomly experience the four intramuscular injection procedures of injectable ARV.
Masking Description: Non applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (24):
- DCBA (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- CDBA (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- DBCA (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- BDCA (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- CBDA (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- BCDA (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- DCAB (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- CDAB (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- DACB (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- ADCB (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- CADB (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- ACDB (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- DBAC (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- BDAC (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- DABC (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- ADBC (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- BADC (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- ABDC (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- CBAD (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- BCAD (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- CABD (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- ACBD (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- BACD (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection
- ABCD (specific order of procedures with type of injection site and/or use virtual reality headset) (Experimental): A: dorsogluteal intramuscular injection, B: ventrogluteal intramuscular injection, C: dorsogluteal intramuscular injection with virtual reality headset, D: ventrogluteal intramuscular injection with virtual reality headset
  Interventions: Procedure: Dorsogluteal intramuscular injection

INTERVENTIONS:
Procedure: Dorsogluteal intramuscular injection — The injection is carried out on the dorsogluteal intramuscular site, without virtual reality headset
  The injection is carried out on the ventrogluteal intramuscular site, without virtual reality headset
  The injection is carried out on the dorsogluteal intramuscular site, with virtual reality headset
  The injection is carried out on the ventrogluteal intramuscular site, with virtual reality headset
  Other Names: Ventrogluteal intramuscular injection; Dorsogluteal intramuscular injection with virtual reality headset; Ventro-gluteal intramuscular injection with virtual reality headset

SUMMARY:
This is a multicenter, randomized, open-label study with a cross-over design. The objective of this project is to compare the intensity of pain induced by injectable antiretroviral (ARV) treatment (Cabotegravir® and Rilpivirine®) in patients infected with HIV-1, depending on the injection site and whether or not they are wearing a virtual reality headset. The reference group being the dorsogluteal injection without headset.

Participants who meet the study criteria will be randomized into 1 of 24 sequences. A sequence is composed by 4 injections procedures: dorsogluteal intramuscular injection (A), ventrogluteal intramuscular injection (B), dorsogluteal intramuscular injection with virtual reality headset (C), ventrogluteal intramuscular injection with virtual reality headset (D).

Each patient will be their own witness and will experience the 4 intramuscular injection procedures of injectable antiretroviral.

The study population are patients carrying HIV-1 and being monitored for this pathology, eligible (naïve patients) or already under Cabotegravir® (CAB) and Rilpivirine® (RPV) injectable treatment.

DETAILED DESCRIPTION:
Five visits will be performed as a standard of care:

Inclusion visit: After checking of the eligibility, patient is informed of the study and an informed note is given. Injection site is examined. If the patient agrees, consent is collected.

Visit D0 (all the patients): examination of the injection zone by the nurse, collection of concomitant treatments (only analgesics and anti-inflammatory drugs) taken by the patient, CAB+RPV injections according to the randomization arm, completion of the numerical scale by the patient following ARV injections, submission of the patient log for the assessment of pain by the patient during the 7 days following the ARV injections.

Follow-up visits (M1, M3, M5 for naïve patients and M2, M4, M6 for treatment-experienced patients): recovery of the patient log with assessment of pain on previous injection, collection of concomitants treatments and adverse events, examination of the injection site by the nurse, injection according the randomization arm, completion of the numerical scale by the patient following the injections, delivery of a new patient note.

End of study visit: recovery of the patient log with assessment of pain on previous injection, collection of concomitants treatments and adverse events, questioning the study procedures, patient's preferred choice between the different injection procedures.

For the research needs,

* The injection site (ventrogluteal and dorsogluteal) will be chosen, by randomisation
* Wearing a virtual reality headset A patient log to assess pain, using a numerical scale (1 to 10), will be filled out by the patient

ELIGIBILITY:
Inclusion Criteria:

* Patient aged at least 18 years;
* Patient infected with HIV-1;
* Patient virologically controlled (VL < 50 copies/ml);
* Patient scheduled to receive treatment with cabotegravir and rilpivirine (naïve patients) or currently on injectable cabotegravir and rilpivirine, prescribed by their referring physician.

Exclusion Criteria:

* Patient(s) on another injectable antiretroviral treatment;
* Patient participating in another clinical trial with medication;
* Patient(s) with epilepsy;
* Patient on antidepressant treatment;
* Patient(s) with psychiatric or behavioral disorders;
* Patient(s) with a history of dizziness and motion sickness that prevents the use of virtual reality headset;
* Patient(s) with visual and hearing impairments that prevent the use of virtual reality headset;
* Patient(s) deprived of liberty, under guardianship or under curatorship;
* Patient(s) not affiliated with a social security scheme;
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-07-24 (Estimated); Study Completion 2026-09-24 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain induced by injectable ARV (Cabotegravir and Rilpivirine) in patients infected with HIV-1, depending on the injection site and whether or not a virtual reality headset is used. | The pain will be self-assessed immediately after the injection, 6-8 hours after the injection, and once a day for the following seven days.
  Composite criterion integrating the measurement of immediate and remote post-injection pain (within 7 days following antiretroviral injections) using a numerical scale from 0 to 10, with immediate post-injection measurement, a second measurement on the first day 6-8 hours after injection then a daily measurement for 7 days.
  The composite criterion will aim to consider pain globally, that is to say all the measurements over 7 days. It is therefore based on the area under the curve of the pain measurement points, normalized by the number of measurement days. This helps increase the first day pain weight, which includes 2 measurements. In practice, this amounts to the sum of the pain measurements (up to 8 measurements in total in absence of missing data), divided by the number of days of measurement (up to 7 days, in the absence of missing data).

SECONDARY OUTCOMES:
Detect the influence of sex on the perception of pain induced by antiretroviral injection. | immediately after the injection; 6-8 hours after the injection; every day for 7 days; at the last visit for each patient (at 7-8 months after inclusion)
  Measurement of post-injection pain (immediate and remote) with one VAS scale (from 0 to 10 with 10 being the worst score) between different patients under dorsogluteal or ventrogluteal with or without virtual reality headset depending on sex
Detect the influence of age on the perception of pain induced by antiretroviral injection. | immediately after the injection; 6-8 hours after the injection; every day for 7 days; at the last visit for each patient (at 7-8 months after inclusion)
  Measurement of post-injection pain (immediate and remote) with one VAS scale (from 0 to 10 with 10 being the worst score) between different patients under dorsogluteal or ventrogluteal with or without virtual reality headset depending on age
Detect the influence of BMI on the perception of pain induced by antiretroviral injection. | immediately after the injection; 6-8 hours after the injection; every day for 7 days; at the last visit for each patient (at 7-8 months after inclusion)
  Measurement of post-injection pain (immediate and remote) with one VAS scale (from 0 to 10 with 10 being the worst score) between different patients under dorsogluteal or ventrogluteal with or without virtual reality headset depending on BMI
Detect the influence of number of injections on the perception of pain induced by antiretroviral injection. | immediately after the injection; 6-8 hours after the injection; every day for 7 days; at the last visit for each patient (at 7-8 months after inclusion)
  Measurement of post-injection pain (immediate and remote) with one VAS scale (from 0 to 10 with 10 being the worst score) between different patients under dorsogluteal or ventrogluteal with or without virtual reality headset depending on number of injections
Compare treatment tolerance depending on the injection site and whether or not a virtual reality headset is worn. The reference group being the dorsogluteal injection without headset | immediately after the injection; 6-8 hours after the injection; every day for 7 days; at the last visit for each patient (at 7-8 months after inclusion)
  Compare all adverse events depending on the injection site and whether or not a virtual reality headset is worn. The reference group being the dorsogluteal injection without headset
Evaluate the representativeness of the cohort of patients treated with injectables, compared to all patients treated for HIV, particularly in terms of gender and ethnic origins, in order to identify indication biases | immediately after the injection; 6-8 hours after the injection; every day for 7 days; at the last visit for each patient (at 7-8 months after inclusion)
  Evaluate the representativeness of the cohort of patients treated with injectables, compared to all patients treated for HIV. Proportion of different ethnic origins and different genders in patients to identify indication biases
Evaluate the satisfaction of the professionals who will perform the injections with a questionnaire | at the last visit for each patient (at 7-8 months after inclusion)
  Evaluate the satisfaction of the professionals who will perform the injections : two questions one on preference (preferred procedure per nurse : A or B or C or D) and one on number (number of procedures per nurse).
Evaluate patient satisfaction about injection procedures with questionnaire | at the last visit for each patient (at 7-8 months after inclusion)
  Evaluate patient satisfaction with injection procedures : one question (which procedure patient prefers : A or B or C or D)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela PIRES ROTEIA, Principal Investigator — CHU Orléans
Locations (5):
- France (5):
  - Center Hospitalier Universitaire d'Orléans, Orléans, Loiret
  - CHD Vendée, La Roche-sur-Yon
  - CH Chartres, Le Coudray
  - CHU Nantes, Nantes
  - CHU Poitiers, Poitiers

REFERENCES:
- [Result] Jonsson-Oldenbuttel C, Ghosn J, van der Valk M, Florence E, Vera F, De Wit S, Rami A, Bonnet F, Hocqueloux L, Hove K, Ait-Khaled M, DeMoor R, Bontempo G, Latham CL, Gutner CA, Iyer S, Gill M, Czarnogorski M, D'Amico R, van Wyk J. Safety and Effectiveness From the Cabotegravir and Rilpivirine Implementation Study in European Locations Study: Phase 3b Hybrid Type III Implementation Study Integrating Cabotegravir + Rilpivirine Long-Acting Into European Clinical Settings. J Acquir Immune Defic Syndr. 2024 Aug 15;96(5):472-480. doi: 10.1097/QAI.0000000000003448. Epub 2024 Jul 9. PMID 38985445
- [Result] Larkin TA, Ashcroft E, Elgellaie A, Hickey BA. Ventrogluteal versus dorsogluteal site selection: A cross-sectional study of muscle and subcutaneous fat thicknesses and an algorithm incorporating demographic and anthropometric data to predict injection outcome. Int J Nurs Stud. 2017 Jun;71:1-7. doi: 10.1016/j.ijnurstu.2017.02.017. Epub 2017 Feb 22. PMID 28273627
- [Result] Gao Y, Xu Y, Liu N, Fan L. Effectiveness of virtual reality intervention on reducing the pain, anxiety and fear of needle-related procedures in paediatric patients: A systematic review and meta-analysis. J Adv Nurs. 2023 Jan;79(1):15-30. doi: 10.1111/jan.15473. Epub 2022 Nov 3. PMID 36330583
- [Result] Chuan A, Zhou JJ, Hou RM, Stevens CJ, Bogdanovych A. Virtual reality for acute and chronic pain management in adult patients: a narrative review. Anaesthesia. 2021 May;76(5):695-704. doi: 10.1111/anae.15202. Epub 2020 Jul 27. PMID 32720308
- [Result] Roldan-Chicano MT, Rodriguez-Tello J, Cebrian-Lopez R, Moore JR, Del Mar Garcia-Lopez M. Adverse effects of dorsogluteal intramuscular injection versus ventrogluteal intramuscular injection: A systematic review and meta-analysis. Nurs Open. 2023 Sep;10(9):5975-5988. doi: 10.1002/nop2.1902. Epub 2023 Jul 14. PMID 37452553
- [Result] Larkin TA, Ashcroft E, Hickey BA, Elgellaie A. Influence of gender, BMI and body shape on theoretical injection outcome at the ventrogluteal and dorsogluteal sites. J Clin Nurs. 2018 Jan;27(1-2):e242-e250. doi: 10.1111/jocn.13923. Epub 2017 Nov 20. PMID 28618093